CLINICAL TRIAL: NCT00159796
Title: A Phase III, Randomized, Placebo-Controlled, Double-Blind Trial Evaluating the Safety and Efficacy of Sublingual Asenapine vs. Olanzapine and Placebo in In-Patients With an Acute Manic Episode Clinical Trial Protocol 7501005 (Secondary Title: ARES)
Brief Title: 3-week Study of Asenapine, Olanzapine and Placebo for Treatment of Bipolar Mania (P07009)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P07009; A7501005 (Other: Schering-Plough)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — asenapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): Asenapine
  Interventions: Drug: Asenapine
- Arm 2 (Active Comparator): Olanzapine
  Interventions: Drug: Olanzapine
- Arm 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asenapine — Asenapine, 3 weeks
  Other Names: Org 5222
  Arms: Arm 1
Drug: Olanzapine — Olanzapine, 3 weeks
  Arms: Arm 2
Drug: Placebo — placebo, 3 weeks
  Arms: Arm 3

SUMMARY:
Bipolar disorder is characterized by mood swings that range from high (manic) to low (depressed) states. Sometimes, symptoms of both depression and mania are present (mixed episodes). Asenapine is an investigational medication for the treatment of manic or mixed episodes of bipolar disorder. This is a 3-week study that will test the safety and efficacy of this medication. Participants will receive either asenapine, olanzapine (a medication that is already approved for the treatment of bipolar mania), or placebo (no active medication). Participants will be required to stay in the hospital for at least the first seven days of treatment. Participants who complete the 3 week study may be eligible to continue in extension studies for an additional 9 (study A7501006) to 49 (study A7501007) weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) diagnosis of bipolar I disorder, current episode manic or mixed.

Exclusion Criteria:

* Participants with unstable medical conditions or clinically significant laboratory abnormalities or participants who are rapid cyclers (i.e., have had 4 or more (including current) mood episodes in the past 12 months); have any other psychiatric disorder other than bipolar I disorder as a primary diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2004-12-14 (Actual); Primary Completion 2006-03-28 (Actual); Study Completion 2006-04-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Day 21 on the Young Mania Rating Scale (YMRS) Total Score | Baseline to Day 21

SECONDARY OUTCOMES:
Change from Baseline to Day 21 in the Clinical Global Impression Scale for use in Bipolar Disorder (CGI-BP) Severity of Mania | Baseline to Day 21
Change from Baseline to Day 21 in the Positive and Negative Symptom Scale (PANSS) Total Score | Baseline to Day 21
Change from Baseline to Day 21 in Montgomery Asberg Depression Rating Scale (MADRS) Total Score | Baseline to Day 21
Readiness for Discharge Questionnaire (RDQ) | Baseline to Day 21
Change from Baseline to Day 21 in Central Nervous System (CNS) Vital Signs | Baseline to Day 21
Change from Baseline to Day 21 in Short Form-36 (SF-36) - Physical Component Summary Scores | Baseline to Day 21
Change from Baseline to Day 21 in the Severity of Extrapyramidal Symptoms (EPS) | Baseline to Day 21
Concomitant Medication Usage | Up to Day 21
Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 30 days after last dose (Up to approximately 51 days)
Change from Baseline to Each Time Point in YMRS Total Score | Days 2, 4, 7, 14, and 21
Change from Baseline to Day 21 in the CGI-BP Severity of Depression | Baseline to Day 21
Change from Baseline to Day 21 in the CGI-BP Severity of Overall Bipolar Illness | Baseline to Day 21
Change from Baseline to Day 21 in SF-36 - Mental Component Summary Scores | Baseline to Day 21
Treatment Satisfaction Questionnaire for Medicine (TSQM) Overall Impact Domain Score at Day 21 | Day 21
Mean Change from Baseline for Vital Signs | Baseline up to Day 21
Change from Baseline to Day 21 in Body Weight | Baseline to Day 21
Summary of Post-Baseline Markedly Abnormal Biochemistry Laboratory Changes/Values | Up to Day 21
Summary of Post-Baseline Markedly Abnormal Endocrinology/Miscellaneous Laboratory Changes/Values | Up to Day 21
Summary of Post-Baseline Markedly Abnormal Metabolic Chemistry Laboratory Changes/Values | Up to Day 21
Summary of Post-Baseline Markedly Abnormal Hematology Laboratory Values | Up to Day 21
Pharmacokinetics - Plasma asenapine concentrations | Day 1 (pre-dose), 7, 14 and 21 (or endpoint)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Suppes T, Eberhard J, Lemming O, Young AH, McIntyre RS. Anxiety, irritability, and agitation as indicators of bipolar mania with depressive symptoms: a post hoc analysis of two clinical trials. Int J Bipolar Disord. 2017 Nov 6;5(1):36. doi: 10.1186/s40345-017-0103-7. PMID 29105003
- [Derived] Michalak EE, Guiraud-Diawara A, Sapin C. Asenapine treatment and health-related quality of life in patients experiencing bipolar I disorder with mixed episodes: post-hoc analyses of pivotal trials. Curr Med Res Opin. 2014 Apr;30(4):711-8. doi: 10.1185/03007995.2013.874988. Epub 2014 Jan 10. PMID 24329543
- [Derived] Szegedi A, Zhao J, McIntyre RS. Early improvement as a predictor of acute treatment outcome in manic or mixed episodes in bipolar-1 disorder: a pooled, post hoc analysis from the asenapine development program. J Affect Disord. 2013 Sep 25;150(3):745-52. doi: 10.1016/j.jad.2013.01.024. Epub 2013 Mar 6. PMID 23473546